CLINICAL TRIAL: NCT06941870
Title: Prospective Interventional Study of Effectiveness of Efanesoctocog Alfa Prophylaxis on Synovial Hypertrophy in Patients With Hemophilia A
Brief Title: Efanesoctocog Alfa Prophylaxis in Patients With Hemophilia A With Synovial Hypertrophy
Acronym: SYNOVIIIUS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPS18168; U1111-1311-1701 (Registry Identifier: ICTRP)
Record Dates: First submitted 2025-04-16; First posted 2025-04-24 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Factor VIII Deficiency
MeSH Terms: conditions — Hemophilia A | interventions — BIVV001

STUDY DESIGN:
Intervention Model Description: Phase 3 in Taiwan, Canada and Australia, Phase 4 in US and Japan.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Efanesoctocog Alfa (Experimental): Participants will receive Efanesoctocog Alfa at 50 international unit per kilogram (IU/kg) intravenous (IV) QW
  Interventions: Drug: Efanesoctocog alfa

INTERVENTIONS:
Drug: Efanesoctocog alfa — Pharmaceutical form:Lyophilized powder in a sterile vial that requires reconstitution with sterile water for injection (diluent)-Route of administration:Intravenous
  Other Names: BIVV001; ALTUVIIIO®

SUMMARY:
The objective of the study is to assess the improvement of synovial hypertrophy during the 12 months of efanesoctocog alfa prophylaxis once per week (QW) in joints with existing evidence of synovial hypertrophy in participants with hemophilia A.

The study duration for each participant is approximately 12 months.

ELIGIBILITY:
Inclusion Criteria: Participant is diagnosed with moderate to severe hemophilia A (defined as less than or equal to (≤)5 percent (%) of endogenous FVIII clotting activity) at the time of consent/assent.

Participant is more than or equal to (≥)12 years old at the time of consent/assent.

Participant has existing synovial hypertrophy, defined as at least 1 eligible* joint by the HEAD-US score (Synovitis score: 1 or 2) at the time of consent/assent.

Participant has at least 1 eligible* joint without planned future major orthopedic procedures (example, arthroscopic synovectomy, radioisotopic or chemical synoviorthesis), or major orthopedic procedures in the past 3 months prior to the screening visit (Visit 1).

*An eligible joint is a joint with existing synovial hypertrophy, as defined by a HEAD-US synovitis score of 1 or 2, considering hypertrophic synovium as an indication of the presence of synovitis Participant has received prophylactic treatment with hemophilia prophylaxis prescriptions in the last 12 months prior to the baseline visit (Visit 2).

Participant is capable of understanding the written Informed Consent Form (ICF)/assent form, provides a signed and witnessed written ICF/assent form, and agrees to comply with the protocol requirements.

If male, no contraceptive measures are required for this study.

If female, is not pregnant or breastfeeding, and one of the following conditions applies:

Is a women of nonchildbearing potential (WONCBP) Is a women of childbearing potential (WOCBP) and agrees to use a highly effective contraceptive method, with a failure rate of less than (<)1 percent during the study treatment period (at least until the Week 52/ End of Treatment [EoT] visit).

A WOCBP must have a negative serum pregnancy test at the screening visit (Visit 1) Exclusion Criteria: Participants are excluded from the study if any of the following criteria apply:

Has other associated clotting disorders at the time of consent/assent. Is already under efanesoctocog alfa treatment. Has a current diagnosis of an factor VIII (FVIII) inhibitor, defined as inhibitor titer ≥0.60 BU/mL.

Has ITI within the last 2 years prior to the baseline visit (Visit 2). Has been enrolled in a concurrent clinical interventional study or exposed to other investigational drug(s) within 3 months prior to screening for this study.

Is currently in an institution because of regulatory or legal order (that is, is a prisoner or a patient who is legally institutionalized).

Is not suitable for participation, whatever the reason, as judged by the investigator, including medical or clinical conditions, or patients potentially at risk of noncompliance to study procedures.

Is an employee or family member of the investigator or site personnel. Is involved in a specific situation during study implementation or the course of the study that may raise ethics considerations.

Has hypersensitivity to efanesoctocog alfa or its components or any of its excipients that, in the opinion of the investigator, contraindicates participation in the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2027-10-25 (Estimated); Study Completion 2027-10-25 (Estimated)

PRIMARY OUTCOMES:
Proportion of joints with improvement in the Hemophilia Early Arthropathy Detection with Ultrasound (HEAD-US) synovitis domain score | From Baseline up to Week 52
  HEAD-US scoring system is a simplified ultrasound scanning procedure to image the elbow, knee, and ankle (index joints) and a scoring system based on an additive scale to define the joint status from disease activity and disease damage parameters to evaluate disease progression and monitor the results of treatment.

SECONDARY OUTCOMES:
Change from baseline in the distribution of joint HEAD-US synovitis score | From Baseline up to Week 52
  HEAD-US scoring system is a simplified ultrasound scanning procedure to image the elbow, knee, and ankle (index joints) and a scoring system based on an additive scale to define the joint status from disease activity and disease damage parameters to evaluate disease progression and monitor the results of treatment.
Number of joints with the HEAD-US synovitis domain score that has remained unchanged or worsened | From Baseline up to Week 52
  HEAD-US scoring system is a simplified ultrasound scanning procedure to image the elbow, knee, and ankle (index joints) and a scoring system based on an additive scale to define the joint status from disease activity and disease damage parameters to evaluate disease progression and monitor the results of treatment.
Percentage of joints with the HEAD-US synovitis domain score that has remained unchanged or worsened | From Baseline up to Week 52
  HEAD-US scoring system is a simplified ultrasound scanning procedure to image the elbow, knee, and ankle (index joints) and a scoring system based on an additive scale to define the joint status from disease activity and disease damage parameters to evaluate disease progression and monitor the results of treatment.
Number of index joint type with the HEAD-US synovitis domain score that has improved, remained unchanged, or worsened | From Baseline up to Week 52
  HEAD-US scoring system is a simplified ultrasound scanning procedure to image the elbow, knee, and ankle (index joints) and a scoring system based on an additive scale to define the joint status from disease activity and disease damage parameters to evaluate disease progression and monitor the results of treatment.
Percentage of index joint type with the HEAD-US synovitis domain score that has improved, remained unchanged, or worsened | From Baseline up to Week 52
  HEAD-US scoring system is a simplified ultrasound scanning procedure to image the elbow, knee, and ankle (index joints) and a scoring system based on an additive scale to define the joint status from disease activity and disease damage parameters to evaluate disease progression and monitor the results of treatment.
Number of participants with at least 1 joint with the HEAD-US synovitis domain score that has improved, remained unchanged, or worsened | From Baseline up to Week 52
  HEAD-US scoring system is a simplified ultrasound scanning procedure to image the elbow, knee, and ankle (index joints) and a scoring system based on an additive scale to define the joint status from disease activity and disease damage parameters to evaluate disease progression and monitor the results of treatment.
Percentage of participants with at least 1 joint with the HEAD-US synovitis domain score that has improved, remained unchanged, or worsened | From Baseline up to Week 52
  HEAD-US scoring system is a simplified ultrasound scanning procedure to image the elbow, knee, and ankle (index joints) and a scoring system based on an additive scale to define the joint status from disease activity and disease damage parameters to evaluate disease progression and monitor the results of treatment.
Change from baseline in average HEAD-US synovitis domain score across all index joints | From Baseline up to Week 52
  HEAD-US scoring system is a simplified ultrasound scanning procedure to image the elbow, knee, and ankle (index joints) and a scoring system based on an additive scale to define the joint status from disease activity and disease damage parameters to evaluate disease progression and monitor the results of treatment.
Change from baseline in total/ domain scores of the HEAD-US | From Baseline up to Week 26
  HEAD-US scoring system is a simplified ultrasound scanning procedure to image the elbow, knee, and ankle (index joints) and a scoring system based on an additive scale to define the joint status from disease activity and disease damage parameters to evaluate disease progression and monitor the results of treatment.
Change from baseline in total/domain scores of the HJHS | From Baseline up to Week 26
  HJHS comprises an assessment of specific features, or items, of the 6 index joints and an assessment of global gait. For each of the 6 joints, the following items are scored: swelling (0 to 3), duration of swelling (0 to 1), muscle atrophy (0 to 2), crepitus on motion (0 to 2), flexion loss (0 to 3), extension loss (0 to 3), joint pain (0 to 2), and strength (0 to 4). The maximum score for an individual index joint is 20. Gait is scored from 0 to 4. The maximum HJHS total score is 124, with a higher score indicating worse joint health.
Change from baseline in total/domain scores of the HJHS | From Baseline up to Week 52
  HJHS comprises an assessment of specific features, or items, of the 6 index joints and an assessment of global gait. For each of the 6 joints, the following items are scored: swelling (0 to 3), duration of swelling (0 to 1), muscle atrophy (0 to 2), crepitus on motion (0 to 2), flexion loss (0 to 3), extension loss (0 to 3), joint pain (0 to 2), and strength (0 to 4). The maximum score for an individual index joint is 20. Gait is scored from 0 to 4. The maximum HJHS total score is 124, with a higher score indicating worse joint health.
Change from baseline in total/ domain scores of magnetic resonance imaging (MRI) | From Baseline up to Week 52
  MRI will be used to detect changes in synovial hypertrophy in index joints of participants.
Change from baseline in patient-reported outcome (PRO) | From Baseline up to Week 52
  Change from baseline in PRO will be assessed by the EQ-5D 5-level (EQ-5D-5L), Patient-Reported Outcomes Measurement Information System - Short Form (PROMIS-SF) version 2.0 Pain Intensity 3a, PROMIS-SF version 1.1 Pain Interference 6a, and PROMIS-SF version 2.0 Physical Function 6b.
Patient reported treatment preference and satisfaction | At Week 52
  Patient reported treatment preference and satisfaction will be assessed through surveys and exit interviews.
Change from baseline in annualized bleeding rate (ABR) (spontaneous, traumatic) | At Week 52
  The ABR will be defined as (number of bleeding episodes occurring during the treatment period)/(duration of the treatment period [days]) × 365.25.
Change from baseline in annualized joint bleeding rate (AjBR) (spontaneous, traumatic) | At Week 52
  The AjBR will be defined as (number of joint bleeding episodes occurring during the treatment period)/(duration of the treatment period [days]) × 365.25.
Change from baseline in target joint resolution, recurrence, or development | At Week 52
  Change from baseline in target joint resolution, recurrence, or development will be assessed.
The occurrence of Adverse Events (AEs), all AEs leading to treatment discontinuation, Serious Adverse Events (SAEs), and Adverse Event of Special Interest (AESIs) | Up to Week 52
  The safety and tolerability of efanesoctocog alfa evaluated in all participants

CONTACTS AND LOCATIONS:
Locations (13):
- United States (4):
  - Orthopedic Institute for Children- Site Number : 8400009, Los Angeles, California
  - Innovative Hematology, Inc.- Site Number : 8400006, Indianapolis, Indiana
  - University of Iowa- Site Number : 8400004, Iowa City, Iowa
  - Ohio State University Hospital East- Site Number : 8400001, Columbus, Ohio
- Canada (2):
  - Investigational Site Number : 1240003, Hamilton, Ontario
  - Investigational Site Number : 1240004, Hamilton, Ontario
- Japan (4):
  - Investigational Site Number : 3920003, Kawasaki, Kanagawa
  - Investigational Site Number : 3920002, Hiroshima
  - Investigational Site Number : 3920001, Saitama
  - Investigational Site Number : 3920004, Tokyo
- Taiwan (3):
  - Investigational Site Number : 1580003, Kaohsiung City
  - Investigational Site Number : 1580001, Taichung
  - Investigational Site Number : 1580002, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: LPS18168 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26646&tenant=MT_SNY_9011